CLINICAL TRIAL: NCT02571803
Title: The Effect of Strict Dietary Intervention on Atherosclerotic Lesions in Patients Diagnosed With Coronary Artery Disease, Assessed by Coronary Computed Tomography Angiography (CCTA).
Brief Title: Dietary Intervention to Stop COronary Atherosclerosis in Computed Tomography
Acronym: DISCO-CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Cezary Kepka, Ass. Prof., National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.15/III/15
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; atherosclerosis; DASH diet
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary And Lifestyle Counseling (Experimental): Patients receiving strict dietary counseling (implementation of the DASH diet) and lifestyle changes support atop of optimal medical treatment as per 2013 ESC guidelines on the management of stable coronary artery disease.
  Interventions: Behavioral: Dietary And Lifestyle Counseling; Other: Optimal Medical Treatment
- Optimal Medical Treatment (Active Comparator): Patients receiving optimal medical treatment as per 2013 ESC guidelines on the management of stable coronary artery disease.
  Interventions: Other: Optimal Medical Treatment

INTERVENTIONS:
Behavioral: Dietary And Lifestyle Counseling — The DASH (Dietary Approaches to Stop Hypertension) diet is a dietary pattern of proven effect on arterial blood pressure reduction. It is rich in fruits, vegetables, whole grains, and low-fat dairy foods; includes meat, fish, poultry, nuts, and beans; and is limited in sugar-sweetened foods and beverages, red meat, and added fats. Dietary counseling will be provided during each of 7 control visits within the 12-month time of observation.
  Other Names: DASH diet implementation with lifestyle changes support
  Arms: Dietary And Lifestyle Counseling
Other: Optimal Medical Treatment — Optimal Medical Treatment as per 2013 ESC Guidelines on the Management of Stable Coronary Artery Disease.
  Other Names: OMT

SUMMARY:
The aim of the study is to determine, wheather strict dietary intervention with the use of the DASH diet atop of optimal medical treatment reduces previously diagnosed coronary atherosclerotic lesions assessed witch coronary computed tomography.

DETAILED DESCRIPTION:
A total of 180 patients with coronary atheroslerotc lesions confirmed in coronary computed tomography (CCT) will be analyzed in a 12-month observation time. Patients will be randomized to two groups in a 1:1 fashion. 1 - optimal medical treatment, 2 - strict dietary intervention with implementation of the DASH diet atop of optimal medical treatment. CCT scans will be performed at screening and at 12 months after randomization. Computed tomography imaging data describing atheroslerotic lesions will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* coronary atheroslerotic lesions confirmed in the screening CCTA with reduction of the artery diameter less than 70% in 2 or more coronary artery segments
* no indications for coronary angiography / revascularization (no documented significant ischemia of myocardium)
* free and informed consent of the person concerned
* willingness to follow the strict directions given by the investigators

Exclusion Criteria:

* any valvular heart disease requiring cardiac surgery (or expected cardiac surgery intervention within 12 moths)
* diagnosis of dilated / hypertrophic cardiomyopathy
* diagnosis of DM t. 2
* past CABG procedure
* women in reproductive age
* known genetic factors with a possible impact on the progres of coronary atherosclerotic lesions (e. i. congenital metabolic disorders, familial hyperlipidemias)
* low quality of the CCTA data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-06 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Percent Of Patheroma Volume (PAV) | 12 months
  Reduction of percent atheroma volume (PAV) measured between baseline and follow-up CT scans.

SECONDARY OUTCOMES:
Pericardial Fat Distribution | 12 months
  Change in pericardial fat distribution between baseline and follow-up CT scans.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Henzel, MD, Study Director — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, Warsaw, Poland

REFERENCES:
- [Derived] Henzel J, Kepka C, Kruk M, Makarewicz-Wujec M, Wardziak L, Trochimiuk P, Dzielinska Z, Demkow M. High-Risk Coronary Plaque Regression After Intensive Lifestyle Intervention in Nonobstructive Coronary Disease: A Randomized Study. JACC Cardiovasc Imaging. 2021 Jun;14(6):1192-1202. doi: 10.1016/j.jcmg.2020.10.019. Epub 2020 Dec 16. PMID 33341413
- [Derived] Makarewicz-Wujec M, Henzel J, Kruk M, Kepka C, Wardziak L, Trochimiuk P, Parzonko A, Demkow M, Kozlowska-Wojciechowska M. DASH diet decreases CXCL4 plasma concentration in patients diagnosed with coronary atherosclerotic lesions. Nutr Metab Cardiovasc Dis. 2020 Jan 3;30(1):56-59. doi: 10.1016/j.numecd.2019.07.013. Epub 2019 Jul 24. PMID 31558416